CLINICAL TRIAL: NCT01105689
Title: Utility of the Urine Calcium Creatinine Ratio as a Screening Tool for Vitamin D Deficiency in Infants and Toddlers
Brief Title: Utility of a Urine Screening Tool for Vitamin D Deficiency in Infants and Toddlers
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Robert Olney, MD, Nemours Children's Clinic
Other Study IDs: 09-171
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Vitamin D Deficiency
Keywords: Urine Calcium to Creatinine Ratio; Hypocalciuria; Infants; Toddlers
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole Blood will be obtained from which we will collect serum and fresh urine which will be used for study labs. Urine and serum may be stored for future studies.
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Vitamin D plays a key role in calcium absorption in the gut and in skeletal development. Vitamin D deficiency is common, affecting an estimated one billion people worldwide, including developed countries. Vitamin D deficiency causes rickets, the most common non-communicable disease of childhood. Rickets causes poor growth and skeletal deformities and, at its most severe, seizures and death. Recent data suggest that children with rickets have an increased risk for developing diabetes mellitus.

Screening for vitamin D deficiency is not commonly done. It is generally diagnosed only after symptoms of rickets have developed. Prevention and treatment is simple and inexpensive. Hence, early detection of vitamin D deficiency through screening would be beneficial. Studies are urgently needed to validate such screening tests.

Calcium balance is tightly regulated in the body and calcium loss in the urine (measured by the urine calcium-to-creatinine ratio) is a sensitive indicator of reduced calcium absorption, such as in vitamin D deficiency.

Objective and Hypotheses. The objective of this study is to evaluate the urine calcium-to-creatinine ratio as a noninvasive and inexpensive screening test for vitamin D deficiency. Our hypotheses are 1) that the urine calcium-to-creatinine ratio correlates with blood vitamin D levels in infants and toddlers at risk for vitamin D deficiency and 2) that this test can be used to screen for vitamin D deficiency.

Potential Impact. A validated screening tool would allow for the detection of vitamin D deficiency before the development of rickets, decreasing the morbidity and mortality of this common disease.

DETAILED DESCRIPTION:
Background:

Insufficient circulating levels of vitamin D is a common problem in both developed and developing countries; it is estimated that over one billion people have vitamin D deficiency at this time. In children, vitamin D deficiency leads to nutritional rickets, which is considered the most common non-communicable disease of children worldwide. Rickets causes significant short term morbidity and mortality through hypocalcemic tetany and seizures, as well as long term morbidity from growth delay and skeletal deformities. Recent data also suggest that children who have had nutritional rickets are three times more likely to develop type 1 diabetes.

There is wide agreement that screening for vitamin D deficiency would be highly beneficial. However, there is debate on how best to do this. Most screening efforts have included serum levels of 25-hydroxy-vitamin D and parathyroid hormone (PTH). However, these assays are complex and are neither available nor affordable for many of the most vulnerable populations.

Calcium excretion in the kidney is a tightly regulated process involving metabolites of vitamin D and PTH. Renal calcium excretion, in the absence of primary renal or parathyroid gland disease, is a sensitive indicator of total body calcium balance. We have shown that renal calcium excretion correlates with blood levels of 25-hydroxy-vitamin D levels in older children and urine calcium-to-creatinine ratios have been shown to distinguish children with active rickets from healthy controls in one Nigerian study. This biomarker is noninvasive and the assays are straight forward and inexpensive. We believe that the urine calcium-to-creatinine ratio has excellent potential as a screening tool for vitamin D deficiency.

Objective and Hypotheses. The objective of this study is to evaluate the urine calcium-to-creatinine ratio as a biomarker of vitamin D deficiency. Our hypotheses are 1) that urine calcium-to-creatinine ratio correlates with serum 25-hydroxy vitamin D level in infants and toddlers at risk for vitamin D deficiency and 2) that the urine calcium-to-creatinine ratio can be used to screen children for vitamin D deficiency. These hypotheses will be tested through two specific aims. Specific Aim 1 is to determine the correlation between the urine calcium-to-creatinine ratio with 25-hydroxy vitamin D levels and with biomarkers of rickets in infants and toddlers at increased risk for vitamin D deficiency. Specific Aim 2 is to determine the sensitivity, specificity, and positive and negative predictive values of one random urine calcium-to-creatinine ratio in relation to biochemical evidence of vitamin D deficiency.

Design. This will be an observational study of infants and toddlers at increased risk for vitamin D deficiency. We will recruit 150 healthy children, 6 to 36 months of age, with risk factors for vitamin D deficiency (premature birth, breast feeding, dairy product avoidance, etc.). Based on previous studies in the US, we anticipate about 12% of these subjects will have vitamin D deficiency. Subjects will have a physical exam targeted to signs of rickets. Laboratories will include a random urine sample for calcium-to-creatinine ratio and blood for calcium, creatinine, alkaline phosphatase, phosphorus, magnesium, intact PTH, and 25-hydroxy vitamin D. Subjects with biochemical evidence of rickets will have x-rays done of the left wrist and knees that will be scored according to previously published rickets scores.

Potential Impact. Vitamin D deficiency is increasingly recognized as a common source of morbidity in both developed and undeveloped countries. The validation of a noninvasive and inexpensive screening tool for vitamin D deficiency would allow for large scale screening of at risk populations and detect this problem early, preventing the morbidities of rickets.

ELIGIBILITY:
Inclusion Criteria:

* In one of the 6 high-risk groups between the age of 6 months and 3 years.

Exclusion Criteria:

* known familial rickets (hypophosphatemic or vitamin D resistant)
* known parathyroid hormone problems
* any child on diuretics
* presence of a chronic disease or use of medications known to affect vitamin D metabolism
* renal insufficiency
* known malabsorption
* rickets secondary to other syndromes (e.g. Fanconi syndrome)

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and Toddlers from 6 months to 3 years part of a group known to be in at least one high-risk group for vitamin D deficiency:
  1. child has been exclusively breast fedfor at least 1 month
  2. darkly pigmented children
  3. children born at a gestational age of 32 weeks or less
  4. recent immigrant from developed country
  5. child is underweight (wt/ht < 10%)
  6. children with bowed legs or wrist enlargement
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olney, MD, Principal Investigator — Nemours Children's Clinic; Matthew Benson, MD, Study Director — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Olney RC, Mazur JM, Pike LM, Froyen MK, Ramirez-Garnica G, Loveless EA, Mandel DM, Hahn GA, Neal KM, Cummings RJ. Healthy children with frequent fractures: how much evaluation is needed? Pediatrics. 2008 May;121(5):890-7. doi: 10.1542/peds.2007-2079. PMID 18450891
- [Background] Gordon CM, Feldman HA, Sinclair L, Williams AL, Kleinman PK, Perez-Rossello J, Cox JE. Prevalence of vitamin D deficiency among healthy infants and toddlers. Arch Pediatr Adolesc Med. 2008 Jun;162(6):505-12. doi: 10.1001/archpedi.162.6.505. PMID 18524739
- [Background] Thacher TD, Fischer PR, Pettifor JM, Lawson JO, Manaster BJ, Reading JC. Radiographic scoring method for the assessment of the severity of nutritional rickets. J Trop Pediatr. 2000 Jun;46(3):132-9. doi: 10.1093/tropej/46.3.132. PMID 10893912
- [Background] Thacher TD, Fischer PR, Pettifor JM, Lawson JO, Isichei CO, Chan GM. Case-control study of factors associated with nutritional rickets in Nigerian children. J Pediatr. 2000 Sep;137(3):367-73. doi: 10.1067/mpd.2000.107527. PMID 10969262
- [Background] Thacher TD, Fischer PR, Pettifor JM. The usefulness of clinical features to identify active rickets. Ann Trop Paediatr. 2002 Sep;22(3):229-37. doi: 10.1179/027249302125001525. PMID 12369487